CLINICAL TRIAL: NCT06854770
Title: The Outreach Project: a Study of Women-led, Trauma Informed Outreach to Foster Equity
Brief Title: STRENGTH Pilot Project: a Study of a Women-led, Trauma-informed Model of Outreach to Foster Equity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Inner-City Women's Initiatives Society (Unknown); Vancouver Foundation (Other)
Responsible Party: Principal Investigator, Victoria Bungay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H18-00069; H18-00069 (Other: UBC Behavioural Research Ethics Board)
Record Dates: First submitted 2025-02-14; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Access to Health Care; Gender-Based Violence; Safety; Access to Social Services; Outreach Intervention
Keywords: pilot study; acceptability study; feasibility study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- STRENGTH Outreach Intervention (Experimental): Participants enrolled in STRENGTH intervention elements
  Interventions: Behavioral: STRENGTH Outreach Intervention

INTERVENTIONS:
Behavioral: STRENGTH Outreach Intervention — The STRENGTH outreach intervention is a community-led, strengths-based, and trauma- and violence-informed program to support self-identifying women who experience interpersonal and structural gender-based violence. The outreach intervention aims to support individuals to achieve self-identified priorities.

SUMMARY:
The goal of this pilot study is to identify the core elements of outreach practice necessary to engage with women experiencing street-involvement who are underserved within health and social care settings. The primary research questions are:

1. How acceptable is the outreach intervention to women experiencing street-involvement?
2. What factors act as barriers or facilitators to acceptability?
3. How feasible is the outreach intervention to enhance women's access to health and social services?

Participants will:

* Meet regularly one-on-one with an outreach worker over an 18-month period
* Co-develop (with the outreach worker) a plan, based on the individuals self-identified needs, for connecting with health and social services
* Be invited to complete surveys at the start of their participation, and again every four months. These surveys ask questions about participants' resiliency, quality of life, independence, safety, and health status
* Be invited to participate in a one-on-one interview with a researcher about their experiences in the study.

DETAILED DESCRIPTION:
The STRENGTH Pilot Project is a community-based, participatory action pilot study to design and test the acceptability of a women-led, trauma and violence informed model of outreach situated in the Downtown Eastside Neighbourhood of Vancouver, British Columbia.

Many women are underserved within health and social care due to numerous environmental factors affecting their access and receipt of services appropriate to their needs. These challenges are shaped by siloed service delivery, isolation, knowledge gaps about services, and negative encounters in support service settings. Outreach activities can build lasting relationships between support workers and women in ways that enhance quality of life and overall wellbeing, and are not harmful or re-traumatizing. The overall aim of the project is to develop and test the acceptability of a model of outreach that is women-led, strengths-based and trauma and violence informed.

In collaboration with community service experts and women with lived experience and drawing on existing empirical evidence concerning outreach interventions as a means to engage underserved women with health and social care, a preliminary model of outreach was developed to be tested within a pilot, single case study design focusing on acceptability of the intervention and feasibility of outreach to enhance women's access to health and social care. Within the intervention, outreach teams work with women in identifying their goals and needs and in partnership, support them to engage with services and supports to address their health and social care service needs.

In this pilot study, we will be evaluating (a) the acceptability of the outreach intervention; (b) environmental factors affecting acceptability; and (c) the feasibility of the intervention to increase women's engagement with appropriate health and social care services.

Because this project is a pilot study, the key research questions being addressed are:

1. How acceptable is the outreach intervention to women experiencing street-involvement?
2. What factors act as barriers or facilitators to acceptability?
3. How feasible is the outreach intervention to enhance women's access to health and social services?

Research activities designed to answer the above research questions include

1. Baseline data collection with women and at 4 month intervals to assess resiliency, quality of life, independence (mastery), safety, and health status;
2. Qualitative interviews with women to study acceptability, satisfaction, burden and appropriateness of the intervention;
3. Chart review of the plan of care documentation to study feasibility of increased engagement with services and women's retention in the intervention;
4. Bi-weekly meetings with outreach workers to identify barriers and facilitators to effective engagement.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a woman, therefore the study is trans-inclusive.
* Have some degree of English proficiency in understanding and communication.
* Live or spend most of their time over a 24-hour period in the Downtown Eastside of Vancouver.
* Age 18 or over.

Exclusion Criteria:

* Women without any degree of English speaking or comprehension proficiency.
* People who self-identify as men.
* Youth under the age of 18.
* Women who do not spend time regularly in the Downtown Eastside of Vancouver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identifying women inclusive of trans women
Enrollment: 37 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Outreach Team Engagement with Individual Participants | From enrollment to end of intervention (up to 18 months)
  Number of times outreach team met with individual participants
Participants' Access to Consistent Health Care | From enrollment to end of intervention (up to 18 months)
  Measured in a binary survey item assessing participants' access to a consistent health care provider
Participants' Confidence in Engaging with Services | From enrollment to end of intervention (up to 18 months)
  Measured in a survey item (self-rated scale from 0-100%) assessing confidence in accessing services

SECONDARY OUTCOMES:
Acceptability of Outreach Intervention | At 12 to 15 months post-enrollment
  Measured using a qualitative interview question: "Are you satisfied with what you achieved in this project?"

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bungay V, Dewar L, Schoening M, Guta A, Leiper W, Jiao S. Co-designing an Outreach Intervention for Women Experiencing Street-Involvement and Gender-Based Violence: Community-Academic Partnerships in Action. Violence Against Women. 2024 Jun;30(8):1760-1782. doi: 10.1177/10778012241233004. Epub 2024 Feb 19. PMID 38374653